CLINICAL TRIAL: NCT00964821
Title: Influenza Specific Humoral and Cellular Immunity After Vaccination in Recipients of Allogeneic and Autologous Hematopoietic Stem Cell Transplantation
Brief Title: Flu Vaccine in Preventing Influenza Infection in Healthy Volunteers and in Patients Who Have Undergone Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 06157; P30CA033572 (NIH); CHNMC-06157; CDR0000652790 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2009-08-22; First posted 2009-08-25 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Nonmalignant Neoplasm
Keywords: stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent childhood large cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent mycosis fungoides/Sezary syndrome; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; aplastic anemia
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neoplasms; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Acute; Leukemia, Hairy Cell; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Anemia, Aplastic | interventions — Influenza Vaccines; Immunoenzyme Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Flu vaccine: Patients and normal volunteers who have received a flu vaccine
  Interventions: Biological: trivalent influenza vaccine; Other: Immunoenzyme technique; Other: Laboratory biomarker analysis
- Non-vaccine: Patients and normal volunteers who have not received the flu vaccine
  Interventions: Other: Immunoenzyme technique; Other: Laboratory biomarker analysis

INTERVENTIONS:
Biological: trivalent influenza vaccine — Patients or normal volunteers who will be vaccinated against the flu.
  Groups: Flu vaccine
Other: Immunoenzyme technique — This test will determine the level of antibodies in participants who have been vaccinated against the flu and those who have not been vaccinated against the flu.
Other: Laboratory biomarker analysis — This test will count the number of T cells (the cells that kill the flu virus) in participants who have been vaccinated against the flu and those who have not been vaccinated against the flu.

SUMMARY:
RATIONALE: Studying immune response to flu vaccine in patients who have undergone a stem cell transplant may help doctors plan the best treatment.

PURPOSE: This clinical trial is studying flu vaccine to see how well it works in preventing infection in patients who have undergone a stem cell transplant and in healthy volunteers.

DETAILED DESCRIPTION:
OBJECTIVES:

* Examine the humoral and cellular memory immune responses to influenza immunization in patients who have undergone autologous or allogeneic hematologic stem cell transplantation.
* Examine the impact of graft-vs-host disease on immune reconstitution and vaccine response in these patients.
* Examine the impact of age ≥ 60 years on immune reconstitution after vaccination in these patients.
* Examine and compare the cellular memory immune response to influenza immunization in healthy volunteers versus the response in these patients.
* Examine the differences between CD8, CD4, and antibody response to circulating flu strains compared to immune response to flu vaccination in immunized vs non-immunized patients who were transplanted at a similar time and from the same transplant source.

OUTLINE: This is a multicenter study. Patients are stratified according to transplantation type and response (allogeneic HCT with no acute or chronic GVHD vs allogeneic HCT with acute or chronic GVHD vs autologous HCT) and patient age (≥ 60 years vs < 60 years).

Beginning 100-364 days post-transplantation patients receive vaccine to immunize against influenza A serotypes specific for influenza seasons 2006-2008, and/or vaccine to immunize against influenza A and B serotypes specific for influenza seasons 2009-2011. Healthy participants receive vaccine to immunize against influenza A serotypes specific for influenza season 2007-2008.

Blood samples from patients and healthy participants are collected at baseline and at days 30, 90, 180, and 360 post-vaccination for humoral immunity and antibody analysis by ELISA and hemagglutination-inhibition test (HAI) testing.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Patient at the City of Hope or Kaiser hospital who underwent prior autologous or allogeneic matched-related hematologic stem cell transplantation (HSCT) or matched-unrelated HSCT for treatment of hematological malignancies, including aplastic anemia or myelodysplastic syndromes

    * Eligible (in accordance with physician's recommendation) to receive the vaccine influenza A serotypes specific for the 2006-2007 or 2007-2008 influenza season
    * Eligible (in accordance with physician's recommendation) to receive the vaccine influenza A or B serotypes specific for the 2009-2010 or 2010-2011 influenza season

      * Patients who are not vaccinated are followed under the study protocol once they are matched to a vaccinated patient on the date of transplant and source of transplant
    * All HLA serotypes allowed
  * Employee volunteer from the City of Hope

    * Meets the requirements for influenza vaccination
    * Eligible to receive the CDC recommended vaccine for influenza A serotypes specific for the 2007-2008 flu season as part of occupational health's vaccination initiative
    * All HLA serotypes allowed

PATIENT CHARACTERISTICS:

* Life expectancy > 9 months
* No HIV seropositivity
* No hepatitis B or C seropositivity

  * Hepatitis B-positive serology by vaccination allowed

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior influenza vaccination after transplantation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stem cell donors, Autologous and Allogeneic HCT patients, Normal volunteers
Sampling Method: Non-Probability Sample
Enrollment: 459 (Actual)
Dates: Start 2007-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Humoral and cellular memory immune responses in patients and healthy volunteers | At Day 0 and 30, 90 and 180 days after vaccine in healthy participants and also at 360 days in transplant patients . 4-5 times in the first 2 years after transplant for transplant patients not vaccinated. One time in normal participants not vaccinated.

SECONDARY OUTCOMES:
Incidence rate of influenza or respiratory incidence in patients after vaccination | 1 year after vaccination or two years after transplant if not vaccinated.
Impact of graft-vs-host disease on immune reconstitution and vaccine response | 1 year after vaccination or two years after transplant if not vaccinated.
Impact of age ≥ 60 years on immune reconstitution of after vaccination | 1 year after vaccination or two years after transplant if not vaccinated.
Differences between antibody and cytokine (CD8 and CD4) response | 180 days after vaccine in healthy participants. 360 days after vaccine in transplant patients. 2 years after transplant for transplant patients not vaccinated. One time in normal participants not vaccinated.

CONTACTS AND LOCATIONS:
Overall Officials: Don Diamond, PhD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope Medical Group, Pasadena, California